## Post Extraction Wound Healing Evaluation of Immediate Complete Denture using IPR Scale

[NCT ID not yet assigned]

**Unique Protocol ID: 01154777474** 

**Document Date: 15/7/2022** 

## **Statistical Analysis:**

Data were presented as means and standard deviation (SD) values. The comparison between any two groups were done using independent t-test (Student's t-test).

Statistical analysis was performed with SPSS 20® (Statistical Package for Social Science) and Microsoft Excel2010. The significant level was set at  $P \le 0.05$ .